CLINICAL TRIAL: NCT02150395
Title: The Impact of Music Therapy on Anxiety in Patients Newly Diagnosed With Cancer & Undergoing Simulation for Radiation Therapy
Brief Title: Impact of Music Therapy on Anxiety in Patients With Cancer Undergoing Simulation for Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 199-13
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Anxiety and Distress
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- music therapy (Experimental): pt received a protocolized music therapy intervention that included altered state induction, music driven guided visualiztion, and psychoeducation on relaxation techniques to be used during simulation for radiation therapy. Prescribed pre-recorded music program provided to be used during simulation.
  Interventions: Other: music therapy
- control (No Intervention): no intervention

INTERVENTIONS:
Other: music therapy
  Arms: music therapy

SUMMARY:
This study looks at the effects of a protocolized music therapy intervention on state anxiety for patients with cancer undergoing simulation for radiation therapy. Simulation, which is an imaging and diagnostic procedure, has been identified as producing significantly high levels of anxiety in many cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with breast cancer, and newly diagnosed patients with head and neck cancer.
* 18 or over.
* Fluent in English.

Exclusion Criteria:

* Under 18 years.
* Pre-existing anxiety disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Reduction in state anxiety | 20 minutes
  pt received a protocolized music therapy intervention that included altered state induction, music driven guided visualiztion, and psychoeducation on relaxation techniques to be used during simulation for radiation therapy. Prescribed pre-recorded music program provided to be used during simulation.

SECONDARY OUTCOMES:
reduced distress | 20 minutes
  pt received a protocolized music therapy intervention that included altered state induction, music driven guided visualiztion, and psychoeducation on relaxation techniques to be used during simulation for radiation therapy. Prescribed pre-recorded music program provided to be used during simulation.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne V Loewy, DA, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States